CLINICAL TRIAL: NCT04581434
Title: Comparative Effectiveness of Trauma-Focused and Non-Trauma-Focused Treatment Strategies for PTSD Among Those With Co-Occurring SUD (COMPASS)
Brief Title: Psychotherapy for PTSD Among Veterans Also Receiving Drug or Alcohol Treatment
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Veterans Research and Education (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #PTSD-2019C1-16009
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Stress Disorders, Post-Traumatic; Substance Use Disorders
Keywords: PTSD; Substance Use Disorders; Psychotherapy; Randomized Clinical Trial; Comparative Effectiveness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma-Focused Therapy (Experimental): Patients randomized to Trauma Focused Therapy will receive either Prolonged Exposure (PE) or Cognitive Processing Therapy (CPT). According to standard VA practice, assignment will be determined according to which trauma-focused therapy the assigned provider is verified to provide; if the assigned therapist is verified in both PE and CPT, the provider will decide which treatment to deliver. PE and CPT are both recommended as frontline treatments by all published PTSD guidelines. The standard treatment length will be 12 weekly sessions; however, patients and providers can collaboratively agree to early completion or extension as warranted.
  Interventions: Behavioral: Prolonged Exposure Therapy; Behavioral: Cognitive Processing Therapy
- Non-Trauma-Focused Therapy (Experimental): Those randomized to non-trauma-focused therapy will receive present centered therapy (PCT). Originally designed as a strong comparator for psychotherapy research that included the components of "good therapy," PCT is now a bona-fide PTSD treatment suggested at the second tier in multiple clinical practice guidelines. The standard treatment length will be 12 weekly sessions; however, patients and providers can collaboratively agree to early completion or extension as warranted.
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Prolonged Exposure Therapy is an individually-delivered treatment for PTSD that includes in vivo exposure to trauma reminders and imaginal exposure to the trauma memory delivered in 90-minute weekly sessions.
  Arms: Trauma-Focused Therapy
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an individually-delivered treatment for PTSD that focuses on challenging and modifying maladaptive beliefs related to the trauma, with an optional written trauma account during weekly 60-minute sessions
  Arms: Trauma-Focused Therapy
Behavioral: Present Centered Therapy — Present Centered Therapy is an individually-delivered treatment for PTSD that focuses on "current life problems as manifestations of PTSD" in weekly 60-minute sessions. It includes psychoeducation and normalization of responses to trauma, problem solving related to current life difficulties and stress identified by patients, and emotional support and validation
  Arms: Non-Trauma-Focused Therapy

SUMMARY:
Many people who have posttraumatic stress disorder (PTSD) also struggle with problematic alcohol or drug use (substance use disorders [SUD]). Patients with both conditions prefer PTSD be treated alongside SUD. However, clinicians don't know if treatments that have been found to help those with PTSD work as well for people who also have SUD. This often leads to delaying PTSD treatment or using psychotherapies without research support. Trauma-focused psychotherapy (TFT) is the type of psychotherapy for PTSD that has been studied most often among people with both PTSD and SUD. It reduces symptoms of PTSD and substance use, although it might not work as well in those who have SUD as those who do not. Further, many patients with both PTSD and SUD do not complete TFT. Another strategy for treating PTSD is non-trauma-focused psychotherapy (NTFT). One NTFT, Present Centered Therapy, has been found to reduce symptoms of PTSD and more patients are able to complete NTFT than are able to finish TFT. However, no one has studied how well Present Centered Therapy works among patients who also have SUD.

We will test which approach (TFT of NTFT) is better for reducing symptoms of PTSD and which is more likely to be completed by patients with both PTSD and SUD at VA healthcare facilities. We will also test to see whether some participants did better than others, so we can learn how to individualize treatment recommendations to patients. Participants will be assigned by chance to either TFT of NTFT. Patients assigned to TFT will receive either Prolonged Exposure or Cognitive Processing Therapy; both are weekly psychotherapies focused on addressing thoughts and/or memories related to their trauma. Those assigned to NTFT will receive Present Centered Therapy, a weekly psychotherapy in which patients learn about how PTSD relates to their current difficulties and problem solve current life difficulties. All participants will also receive SUD treatment. Participants will answer questions about their symptoms and experience with treatment before, right after they finish, and three and six months after they finish PTSD treatment. At the end of the study we will compare which treatment approach worked better to decrease PTSD symptom severity and which treatment patients were better able to complete. We will also track other outcomes that are important to patients (e.g., how they are doing in their relationships).

DETAILED DESCRIPTION:
Background and Significance: Posttraumatic stress disorder (PTSD) and substance use disorder (SUD) comorbidity is common. The Veterans Affairs (VA)/Department of Defense Clinical Practice Guideline for PTSD strongly recommends providing guideline-concurrent care for PTSD alongside SUD treatment, but there is insufficient evidence about which guideline-recommended treatments for PTSD work best in this population. Trauma-focused therapy (TFT) is a frontline treatment approach; yet its effectiveness is less well-established among patients with co-occurring SUD, and TFT dropout rates are uniquely high in this population. Multiple guidelines suggest non-trauma-focused treatment (NTFT) as a second-line treatment approach for PTSD; higher completion rates for some NTFT (e.g., Present Centered Therapy) may make this strategy particularly effective for those with comorbid SUD. Despite providers' desire for an NTFT option for patients with PTSD/SUD, no guideline-recommended NTFTs have been evaluated in those with the comorbidity

Study Aims: Our long-term objective is to improve the lives of patients with co-occurring PTSD and SUD. To meet this objective, we will conduct a pragmatic randomized clinical trial that will yield decisive data regarding the comparative effectiveness of two evidence-based approaches for the treatment of PTSD in this understudied patient population: trauma-focused and non-trauma-focused psychotherapy. The major aims are: (1) Determine whether TFT differs at a clinically-meaningful magnitude from NTFT in its effects on posttreatment PTSD symptoms among patients with co-occurring PTSD and SUD (2) Determine whether patients with co-occurring PTSD and SUD randomized to TFT drop out of PTSD treatment more often than those randomized to NTFT, and (3) Determine if TFT differs at a clinically-meaningful level from NTFT in PTSD symptom reduction and number of PTSD therapy sessions attended in patients with varying (a) levels of baseline SUD severity, (b) classes of misused substances, and (c) treatment preferences.

Study Description: We propose a prospective, pragmatic randomized comparative effectiveness trial at 14 VA Medical Center sites (11 confirmed). Randomization will occur at the patient level and will assign participants to either (1) TFT (Prolonged Exposure or Cognitive Processing Therapy) or 2) NTFT (Present Centered Therapy). All participants will also receive concurrent SUD treatment-as-usual. Participants will complete self-report measures and a clinician-administered interview pretreatment, posttreatment, and six-months posttreatment. 420 participants (210 per arm) will be veterans seeking outpatient SUD treatment in an enrolled clinic who meet DSM-5 criteria for a current SUD and PTSD. The sample will be diverse in sex, race, age, and geography. Main outcomes will be PTSD symptom severity measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5), and PTSD treatment dropout (dichotomous indicator of completion of all PTSD treatment sessions). Major Aim 1 will be tested using a linear mixed model using study intervention, assessment point, and their interaction as fixed effects and including random effects for participant, clinician, and study site. Major Aim 2 will be testing using a random effects logistic regression of therapy retention on intervention and baseline CAPS incorporating random effects for clinician and site.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Initiate an episode of outpatient SUD treatment at an enrolled facility.
2. meet DSM-5 criteria for a current SUD (Tobacco Use Disorder alone is not sufficient for inclusion).
3. Report substance use in the past 30 days (or in the 30 days prior to entering a controlled environment if exiting said controlled environment at time of enrollment)
4. meet DSM-5 criteria for PTSD
5. provide informed consent and be willing to be randomized to PTSD treatment condition
6. agree to not receive non-study, active psychotherapy for PTSD during study treatment

EXCLUSION CRITERIA:

1. Severe cognitive impairment
2. Current suicidal or homicidal intent with a specific plan
3. Unstable psychotic or manic symptoms not attributable to SUD
4. More than 30 days between index outpatient SUD intake/treatment planning appointment & consent or more than 90 days between the index outpatient SUD visit and the first PTSD psychotherapy session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Clinician Administered Scale for PTSD -5 (CAPS-5) Severity Score | Immediately after ending treatment
  PTSD Symptom Severity - Clinician Assessed; range 0-80; higher scores = greater severity.
PTSD Treatment Non-completion | Immediately after ending treatment
  Proportion of veterans who do not complete a full course of assigned PTSD treatment

SECONDARY OUTCOMES:
PTSD Checklist-5 (PCL-5) | Immediately after ending treatment
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms
PTSD Checklist-5 (PCL-5) | 3-months after ending treatment
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms
PTSD Checklist-5 (PCL-5) | 6-months after ending treatment
  PTSD Symptom Severity - Self-Reported; Range = 0-80; higher scores = more severe symptoms
% Days with drug use or heavy drinking over prior 28 days | Immediately after ending treatment
  Substance use as measured by the Timeline Follow-Back Interview (TLFB)
% Days with drug use or heavy drinking over prior 28 days | 3 months after ending treatment
  Substance use as measured by the Timeline Follow-Back Interview (TLFB)
% Days with drug use or heavy drinking over prior 28 days | 6 months after ending treatment
  Substance use as measured by the Timeline Follow-Back Interview (TLFB)
Clinician Administered Scale for PTSD -5 (CAPS-5) Severity Score | 3 months after treatment
  PTSD Symptom Severity - Clinician Assessed; range 0-80; higher scores = greater severity.
Clinician Administered Scale for PTSD -5 (CAPS-5) Severity Score | 6 months after treatment
  PTSD Symptom Severity - Clinician Assessed; range 0-80; higher scores = greater severity.
Short Inventory of Problems, Revised (SIP-R) | Immediately after treatment
  Problems associated with drug or alcohol use; range = 0-51, higher scores = more severe
Short Inventory of Problems, Revised (SIP-R) | 3-months after treatment
  Problems associated with drug or alcohol use; range = 0-51, higher scores = more severe
Short Inventory of Problems, Revised (SIP-R) | 6-months after treatment
  Problems associated with drug or alcohol use; range = 0-51, higher scores = more severe
Brief Inventory of Psychosocial Functioning (BIPF) | Immediately after treatment
  PTSD-related psychosocial functioning; higher scores = more severe
Brief Inventory of Psychosocial Functioning (BIPF) | 3 months after treatment
  PTSD-related psychosocial functioning; higher scores = more severe
Brief Inventory of Psychosocial Functioning (BIPF) | 6 months after treatment
  PTSD-related psychosocial functioning; higher scores = more severe
Insomnia Severity Index | Immediately after treatment
  Self-reported sleep disturbances; range 0-28; higher scores = more severe
Insomnia Severity Index | 3 months after treatment
  Self-reported sleep disturbances; range 0-28; higher scores = more severe
Insomnia Severity Index | 6 months after treatment
  Self-reported sleep disturbances; range 0-28; higher scores = more severe
Dimensions of Anger Reactions (DAR) | Immediately after treatment
  Self-reporter anger; range = 2-25; higher scores = more severe
Dimensions of Anger Reactions (DAR) | 3 months after treatment
  Self-reporter anger; range = 2-25; higher scores = more severe
Dimensions of Anger Reactions (DAR) | 6 months after treatment
  Self-reporter anger; range = 2-25; higher scores = more severe
WHO Quality of Life, Brief (WHOQOL-BREF) | Immediately after treatment
  Self-reported quality of life; higher score = better quality of life
WHO Quality of Life, Brief (WHOQOL-BREF) | 3 months after treatment
  Self-reported quality of life; higher score = better quality of life
WHO Quality of Life, Brief (WHOQOL-BREF) | 6 months after treatment
  Self-reported quality of life; higher score = better quality of life
Patient Health Questionnaire-9 (PHQ-9) | Immediately after treatment
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Patient Health Questionnaire-9 (PHQ-9) | Three months after treatment
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Patient Health Questionnaire-9 (PHQ-9) | Six months after treatment
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Client Satisfaction Questionnaire - 8 (CSQ-8) | Immediately after treatment
  Treatment satisfaction; range = 8-32; higher scores = more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Kehle-Forbes, PhD, Principal Investigator — Minneapolis VA Healthcare System; Hildi Hagedorn, PhD, Principal Investigator — Minneapolis VA Healthcare System
Locations (14):
- United States (14):
  - San Diego VA Healthcare System, San Diego, California
  - Tampa VA Medical Center, Tampa, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Syracuse VA Medical Center, Syracuse, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Cincinnati VA Healthcare System, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Salt Lake City VA Healthcare System, Salt Lake City, Utah
  - Puget Sound VA Healthcare System, Seattle, Washington
  - Madison VA Medical Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ackland PE, Hagedorn HJ, Kenny ME, Salameh HA, Kehle-Forbes SM, Gustavson AM, Karimzadeh LE, Meis LA. Using brief reflections to capture and evaluate end-user engagement: a case example using the COMPASS study. BMC Med Res Methodol. 2024 May 2;24(1):103. doi: 10.1186/s12874-024-02222-5. PMID 38698315
- [Derived] Kehle-Forbes SM, Nelson D, Norman SB, Schnurr PP, Shea MT, Ackland PE, Meis L, Possemato K, Polusny MA, Oslin D, Hamblen JL, Galovski T, Kenny M, Babajide N, Hagedorn H. Comparative effectiveness of trauma-focused and non-trauma-focused psychotherapy for PTSD among veterans with comorbid substance use disorders: Protocol & rationale for a randomized clinical trial. Contemp Clin Trials. 2022 Sep;120:106876. doi: 10.1016/j.cct.2022.106876. Epub 2022 Aug 18. PMID 35987487